CLINICAL TRIAL: NCT03412474
Title: Evaluation of Postoperative Analgesic Effects of Bilateral Suprazygomatic Maxillary Nerve Block Using Bupivacaine and Dexmedetomidine in Children Undergoing Cleft Palate Repair Under General Anesthesia:Randomized Controlled Trial
Brief Title: Suprazygomatic Block in Cleft Palate Surgery in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAGAA AHMED HERDAN, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: suprazygomatic block
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Cleft Palate
Keywords: suprazygomatic block, dexmedetomidine
MeSH Terms: conditions — Cleft Palate | interventions — Bupivacaine; Dexmedetomidine; Acetaminophen

STUDY DESIGN:
Intervention Model Description: comparison of the analgesic effect of adding dexmedetomidine to bupivacaine with the analgesic effect of using bupivacaine alone in bilateral SMB for children undergoing CP repair under general anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be planned that neither the doctors (investigators) nor the patients' guardians or even children themselves will be aware of the group allocation and drug received. The study drugs will be prepared by an anesthesiologist not involved in performing the block, patient care or in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): Patients will receive 0.2 ml/kg/side of bupivacaine (0.125%).
  Interventions: Drug: Bupivacaine; Drug: paracetamol
- Dexmedetomidine (Active Comparator): Patients will receive 0.2 ml/kg/side of bupivacaine (0.125%) + 0.5 µ/kg of dexmedetomidine.
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine; Drug: paracetamol

INTERVENTIONS:
Drug: Bupivacaine — The study drugs will be prepared by an anesthesiologist not involved in performing the block, patient care or in data collection. Patients will be randomly allocated into two groups of 40 patients each:
  Group A: will receive 0.2 ml/kg/side of bupivacaine (0.125%).
Drug: Dexmedetomidine — Group B: will receive 0.2 ml/kg/side of bupivacaine (0.125%) + 0.5 µ/kg of dexmedetomidine.
  Arms: Dexmedetomidine
Drug: paracetamol — paracetamol

SUMMARY:
Cleft palate (CP) is a common congenital malformation, with an incidence ranging from 0.1 to 1.1 per 1000 births depending on the population group (liau et al, 2010). Early surgery is necessary to reduce phonation and feeding difficulties and reduce complications such as frequent sinusitis and other respiratory tract infections (Takemura et al., 2002).

CP repair is painful, necessitating high doses of intravenous (I.V.) opioids. Therefore, the risk of postoperative respiratory depression and airway obstruction is important, and continuous monitoring is required during the initial 48h postoperatively (Roulleau et al, 2003).

Maxillary nerve block using the suprazygomatic approach is used in children since it presents a lower rate of complications (Captier et al, 2009). By this way, one can reach the nerve as it exits the skull at the foramen rotundum within the pterygopalatine fossa, before the location where its nervous branches innervate the palate (Prigge et al, 2014). This simple, reliable and almost risk-free approach can yield an effective and prolonged anesthesia with a clear decreased use of morphine agents during and after cleft lip-palate surgery in small children (Mesnil et al, 2010). The nerve block must be bilateral. The local anesthetic (LA) is directly injected in the middle part of the fossa at a distance from the foramen rotundum to avoid any trauma to the nerve or vascular injury, as soon as the tip of the needle has crossed the temporal muscle (Binet et al, 2015).

Various adjuvants to local anesthetics to increase the duration of block are described in the literature and used in the daily clinical practice. Dexmedetomidine is a selective alpha 2 (α2) adrenergic agonist with both analgesic and sedative properties. Animal studies showed that perineural dexmedetomidine added to bupivacaine or ropivacaine prolongs the duration of sensory and motor block (Brummett et al, 2011). Other clinical studies investigated the use of dexmedetomidine in patients undergoing ulnar nerve, axillary brachial and greater palatine nerve blocks, showed faster onset time and longer duration of block (Marhofer et al, 2013/ Esmaoglu et al, 2010& Obayah et al, 2010).

DETAILED DESCRIPTION:
Preoperative assessment:

The day prior to surgery, all patients will undergo pre-anesthetic checkup including detailed history, physical, systemic examination and weight of the patient. All patients will be investigated for exclusion of any of the above mentioned contraindications. Laboratory work needed will include: Complete Blood Count (CBC); Prothrombin Time and Concentration (PT& PC); Partial Thromboplastin Time (PTT) and Bleeding Time (BT). All children will be kept nil per mouth 6-8 h for solids and 2 h for clear liquids.

Preparation of the patient:

Written consent and emergency resuscitation equipments including airway devices, pediatric advanced life support drugs for LA toxicity will be available.

Intraoperative management:

All patients in this study will be anesthetized by the same team of anesthesiologists and operated upon by the same surgeon who will be unaware of the study medications.

General anesthesia will be standardized for all patients in both groups using 8 MAC sevoflurane in 100% O2 with appropriate size face mask. Intraoperative monitoring will include ECG, pulse oximetry, noninvasive blood pressure, capnography and temperature probe. After intravenous access securing, endotracheal intubation with appropriate size to the patient's age will be performed after administration of 2 mg/kg propofol.

After orotracheal intubation, assisted mechanical ventilation using Ayre's T- piece will be used to maintain end-tidal carbon dioxide at 35±5 mmHg. General anesthesia will be maintained with 2-3 MAC sevoflurane.

Intraoperatively, patients will receive an infusion of normal saline 0.9% solution 4ml/ kg / h.

Bilateral SMB will be performed before surgery in anesthetized children, after aseptic preparation of the skin. The patient will be in supine position with the head in neutral position. The puncture site will be at the frontozygomatic angle, at the junction of the upper edge of the zygomatic arch and the frontal bone. A needle with 50 mm length and 25 gauge will be inserted perpendicular to the skin. It will be advanced to reach the greater wing of sphenoid at approximately 20 mm depth, then withdrawn a few millimeters and will be redirected toward the nasolabial fold in a 20° forward and 10° downward direction. The progression in the pterygopalatine fossa will be 35 to 45 mm. Loss of resistance after passing through the temporalis muscle will assist in determining the puncture depth. After a negative blood aspiration test, 0.2 ml/kg of the blinded study solution will be injected on each side (Captier et al, 2009).

MAP, HR, SPO2 and end-tidal CO2 will be recorded before induction of anesthesia, before block, after the block and every 10 minutes till end of surgery. Skin incision will be made 20 minutes after SMB block. An increase in HR and MAP above 20% of baseline values with skin incision will be considered as a sign of inadequate analgesia. In this case, fentanyl 1 µg/kg will be given intravenously, and the case will be excluded from the study.

Immediate complications related to regional anesthesia will be recorded:

* Systemic toxicity related to local anesthetics (seizures, heart rhythm, or conduction disorder)
* Bleeding at puncture site
* Pupil alteration and ocular lesion

Before the end of surgery, IV paracetamol 15 mg/kg and dexamethasone 0.2 mg/kg will be administered.

After completion of the surgical procedure, extubation will be done after ensuring adequate orogastric suction and patients will be transferred to the postanesthesia care unit (PACU).

In PACU: MAP, HR, modified CHEOPS, POV and sedation score will be recorded on admission to PACU, 1, 4, 8, 12, 18, 24h postoperatively by an observer who will be unaware of the study protocol.

Postoperative pain will be measured using a modified Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) (Taddio et al, 1995).

CHEOPS = SUM (points for all 6 parameters)

Interpretation:

* minimum score: 4
* maximum score: 13 Patients with modified CHEOPS > 6 will be given rescue analgesia with 15 mg/kg paracetamol intravenously. Those with modified CHEOPS of 4-5 will be given paracetamol 25-40 mg/kg as suppository. Pain scores will be recorded every 10 minutes after administration of rescue analgesia to evaluate pain relief or need for further rescue analgesia. The number of children who will need postoperative rescue analgesics and the duration of analgesia that will be taken at the time when an analgesic is required will be recorded.

Postoperative vomiting episodes will be recorded and treated with intravenous metoclopramide 0.5 mg/kg. Postoperative sedation will be assessed using sedation score described by Culebras et al, 2001 (1. Awake and alert. 2. Sleeping but easily arouses to voice or light touch. 3. Arouses to loud voice or shaking. 4. Arouses with painful stimuli only. 5. Unarousable).

Delayed complications of the blocks will be also investigated and recorded as hematoma, restricted mouth opening, vision, sensory or motor deficit, eating disorder, and local infection.

The parents will be asked to evaluate their satisfaction regarding pain control at the end of 48h postoperatively through 5-point Likertscale (1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied).

Patients will be discharged from the hospital when they are pain free and there is no other medical reason to admit them to a surgical ward.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 5 years
* Children scheduled for primary surgery for soft palate cleft or soft and hard palate clefts
* Gender: both

Exclusion Criteria:

* Parent refusal
* History of developmental delay or mental retardation, which will make observational pain intensity assessment difficult
* Hypersensitivity to any local anesthetics
* Bleeding diathesis
* Children with co-morbid conditions like congenital heart disease, respiratory pathology and central nervous system disorders
* Skin lesions or wounds at the puncture site of the proposed block

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
modified Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) | 24 hours
  postoperative pain assessment in children minimum score: 4, maximum score: 13 Patients with modified CHEOPS > 6 will be given rescue analgesia

SECONDARY OUTCOMES:
time to first analgesia | 24 hours
  time of intravenous paracetamol requirment postoperatively
5-point Likert scale | 24 hours
  parent satisfaction score
  (1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No